CLINICAL TRIAL: NCT05047107
Title: Characterising Risk and Biology Of Smouldering Myeloma for Early Detection Of Symptomatic Myeloma
Brief Title: Biology and Genetics of Smouldering Myeloma
Acronym: COSMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 129657
Record Dates: First submitted 2021-09-15; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Smouldering Myeloma; MGUS; Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BM aspirates and blood samples will be processed to extract tumour and non-tumour cells, as well as plasma and sera. Mononuclear cells (MNCs) will be prepared from these samples by centrifugal sedimentation, or red cell lysis, and plasma cells will be selected using immuno-magnetic beads coupled to monoclonal antibody specific to the plasma cell marker, CD138. In some cases, purified MM cells will be isolated by negative selection using RosetteSep method, which depletes immature progenitors, T-lymphocytes and NK cells. Immune cells, including CD4 and CD8 T cells will be separated by similar means for further assessment.
  MM cells, immune cells and bulk MNCs will be frozen and stored for future DNA and RNA extraction. Cell lysates will be made for immuno-blotting and live cells will be frozen for use in functional assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Non-interventional study

SUMMARY:
Observational clinical trial recruiting Smouldering Myeloma patients (SMM) or potential SMM patients. Study involves collecting blood and bone marrow samples to determine the features of the tumour genome and BM microenvironment, including immune dysfunction that are key drivers of progression from precursor conditions (MGUS and SMM) to MM.

DETAILED DESCRIPTION:
MM is a cancer of plasma cells characterised by bone marrow infiltration by malignant plasma cells, kidney impairment, bone pain and elevated calcium levels1. There are approximately 5,500 new cases diagnosed annually in the UK, with a median survival of 5 years2. Significantly, despite improvements in conventional treatment options, MM remains incurable; patients inevitably relapse and will eventually die from their disease.3 MM is always preceded by defined precursor conditions, termed MGUS, and SMM. However, only 7% of MGUS patients and 50% of SMM patients progress to MM over a 5-year period4. In the UK, current practice favours commencing treatment only when there is evidence of end organ damage as the overall benefit of initiating early therapy is uncertain.

There is an increasing understanding that progression is determined by evolving changes in the tumour genome5 and changes in the immune microenvironment which support tumour growth, leading to progressively dysfunctional anti-tumour immunity. This project correlates changes in the tumour genome and immune microenvironment in individual patients with tumour progression and also aims to compare characteristics in patients with good and poor clinical outcomes with the objective of defining the drivers for disease progression. Furthermore, we aim to explore the use of blood samples to monitor tumour dynamics and immune function. Finally, we will also study the spatial distribution of immune cells and tumour cells in the bone marrow.

Clinical impact: A deeper understanding of the pathogenesis of MM will allow us to risk stratify patients with MGUS and SMM, and manage them accordingly as well as identifying subgroups of patients with MM who require different types of therapies, eg. more intensive multi-drug approaches for patients with adverse risk genetics.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with a confirmed or suspected diagnosis of MGUS, SMM, or MM.

Exclusion Criteria:

* Patients under the age of 18
* Patients with active symptomatic myeloma at diagnosis
* Patients with no evidence of MGUS, sMM or MM
* Patients with rapidly rising paraprotein or serum free light chains suggestive of progressive disease at time of diagnosis or inclusion into study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any individual with a confirmed or suspected diagnosis of MGUS, SMM, or MM.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Genomic markers of progression | 5 years
  To characterise genomic markers of progression by sequencing and studying the biology of bone marrow (BM) derived tumour cells.

SECONDARY OUTCOMES:
Immune biomarkers | 5 years
  To define clonal heterogeneity and biomarkers of progression using liquid biopsies(blood), comparing with BM, and exploring the utility of serial samples.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No